CLINICAL TRIAL: NCT04299932
Title: Electroacupuncture for Stress-predominant Mixed Urinary Incontinence: a Three-armed Randomized Controlled Trial
Brief Title: Acupuncture for Stress-predominant Mixed Urinary Incontinence
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Collaborators: Ministry of Science and Technology of the People´s Republic of China (Other Government)
Responsible Party: Principal Investigator, Liu Zhishun, Dean of Acupuncture Department of Guang'anmen Hospital, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019-241-KY
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Mixed Urinary Incontinence
Keywords: acupuncture; stress-predominant mixed urinary incontinence
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Electroacupuncture(EA) group (Experimental): Participants in EA group will receive treatment at bilateral Bladder Meridian (BL) 33 [Zhongliao], BL35 [Huiyang] and Spleen Meridian (SP) 6 [Sanyinjiao]. The EA treatment will last 30mins for each session, 3 sessions a week (ideally every other day) for a succession of 8 weeks.
  Interventions: Procedure: Electroacupuncture
- Sham Electroacupuncture (SA) group (Sham Comparator): Participants in SA group will receive treatment at bilateral sham BL33 [Zhongliao], sham BL35 [Huiyang] and sham SP6 [Sanyinjiao]. The SA treatment will last 30mins for each session, 3 sessions a week (ideally every other day) for a succession of 8 weeks.
  Interventions: Procedure: Sham electroacupuncture
- Waiting List (WL) group (No Intervention): Participants in WL group will be followed up for 20 weeks. Participants only receive healthcare education and advice on lifestyle modification, which will be received by all the participants in the three groups.

INTERVENTIONS:
Procedure: Electroacupuncture — BL33 is located in the third posterior sacral foramen; BL35, 0.5 cun (≈10mm) lateral to the extremity of the coccyx; and SP6 posterior to the medial border of the tibia, 3 cun superior to the prominence of the medial malleolus. BL33 will be inserted by needles of 0.30×75mm size at the angle of 45°, inward and downward, till the depth of 60-70mm. BL35 will be inserted by needles of 0.30×75mm size, slightly outward and upward, till the depth of 60-70mm. SP6 will be inserted by needles of 0.30×40mm till the depth of 25-30mm. All the needles will be lifted, thrust and twisted evenly for three times, right after insertion, to induce the sensation of deqi. Electronic acupuncture apparatus (Yingdi KWD 808 I electro pulse acupuncture therapeutic apparatus, Changzhou Yingdi Electronic Medical Device Co., Ltd) will be connected to the three pairs of needles transversally, with continuous wave of 20 Hertz (Hz), electric current of 2-6.5 milliampere (mA) for BL33 and BL35, and 1mA-3.5mA for SP6.
  Other Names: EA
  Arms: Electroacupuncture(EA) group
Procedure: Sham electroacupuncture — Sham BL33 is in the area of 1 cun (≈20mm) horizontally outside BL33; sham BL35, 1 cun (≈20mm) horizontally outside BL35; Sham SP6, in the middle of SP6 and tendons. The three pairs of acupoints will be inserted by needles of 0.30×40mm size to a depth of 2-3mm till the needles can stand still. No manipulations will be conducted, and the sensation of deqi will not be induced. Electronic acupuncture apparatus (Yingdi KWD 808 I electro pulse acupuncture therapeutic apparatus, Changzhou Yingdi Electronic Medical Device Co., Ltd) will be connected to the three pairs of needles transversally, with continuous wave of 20Hz and minimal electric current (ideally at a degree which participant can just percept). In about 30 seconds, the electric current will be turned down, leaving the indicator light and ticking sound on.
  Other Names: SA
  Arms: Sham Electroacupuncture (SA) group

SUMMARY:
The investigators plan to conduct this multi-center, three-armed, randomized controlled trial to evaluate the efficacy of electroacupuncture (EA), compared with sham electroacupuncture (SA) and waiting list (WL) on participants with stress-predominant mixed urinary incontinence (MUI).

DETAILED DESCRIPTION:
MUI tends to present with more severe symptoms and put greater burden on the health of individual and economy of society. Current European Association of Urology (EAU) guideline on incontinence recommends to initiate treatment targeted at predominant component of MUI. However, as to whether the interventions for stress urinary incontinence (SUI) can be effectively generalized to stress-predominant MUI, there is still no powerful evidence to support it. It is necessary to seek for interventions specific to stress-predominant MUI. Results of previous studies indicated that acupuncture might help to relieve the incontinence symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MUI by the coexistence of SUI and urgency urinary incontinence (UUI) symptoms in accordance with EAU guideline;
2. Female participants aged between 35 and 75;
3. Stress index > urge index in accordance with Medical, Epidemiologic, and Social aspects of Aging(MESA) questionnaire；
4. Symptoms of MUI for at least three months, and stress IEF outnumber 50% total IEF documented in 3-day voiding diary;
5. Less than 12 micturition episodes in average 24 hours documented in 3-day voiding diary;
6. Positive cough stress test;
7. Urine leakage > 1 g in 1-hour pad test;
8. Voluntary participation in the trial and signed written informed content.

Exclusion Criteria:

1. Urgency-predominant MUI, pure SUI, pure UUI, overflow urinary incontinence (UI) and neurogenic bladder;
2. Uncontrolled symptomatic urinary tack infection;
3. Tumor in urinary system and pelvic organ;
4. Pelvic organ prolapse ≥ degree Ⅱ；
5. Residual urine volume ≥ 100ml；
6. History of treatments targeted at UI, such as acupuncture, PFMT and medications in the previous one month;
7. History of surgery targeted at UI or in pelvic floor, including hysterectomy;
8. Uncontrolled diabetes or severe high blood pressure;
9. Nervous system diseases that may hamper the function of urinary system, such as Multiple sclerosis, Alzheimer's disease, Parkinson's disease, spinal cord injury, cauda equina nerve injury, or multiple system atrophy;
10. Severe heart, lung, brain, liver, kidney, mental illness, coagulation dysfunction or with obvious cognitive dysfunction
11. Installed cardiac pacemaker;
12. Inconvenient or unable to walk, run, go up and down stairs;
13. Allergy to metal, severely fear of acupuncture needles or unbearable to EA;
14. Pregnant at present, plan to conceive in future one year, at lactation period or within 12 months after childbirth.

Ages: 35 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 232 (Estimated)
Dates: Start 2020-10-09 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with at least 50% reduction of mean 24-hour stress incontinence episode frequency (IEF) from baseline. | week 8
  The stress IEF will be documented in 3-day voiding diary.

SECONDARY OUTCOMES:
Proportion of participants with at least 50% reduction of urinary leakage amount from baseline. | week 8
  The urinary leakage amount will be measured by 1 hour pad test.
Change of urinary leakage amount from baseline | week 8
  The urinary leakage amount will be measured by 1 hour pad test.
Proportion of participants with at least 50% reduction of mean 24-hour stress IEF from baseline. | week 4，week 20 and week 32
  The stress IEF will be documented in 3-day voiding diary.
Change of mean 24-hour IEF from baseline. | week 4，week 8, week 20 and week 32.
  The IEF will be documented in 3-day voiding diary.
Change of mean 24-hour stress IEF from baseline | week 4，week 8, week 20 and week 32.
  The stress IEF is documented in 3-day voiding diary.
Proportion of participants with at least 50% reduction of mean 24-hour IEF from baseline | week 4，week 8, week 20 and week 32
  The IEF will be documented in 3-day voiding diary.
Change of total and sub-score of International Consultation on Incontinence Questionnaire-short form (ICIQ-SF) from baseline. | week 4，week 8, week 20 and week 32
  ICIQ-SF questionnaire is a validated questionnaire to assess the severity of incontinence symptoms and influence on QoL in the past four weeks. The questionnaire includes items of IEF, urinary leakage amount and general influence on life to be scored. Total number of the score ranges from 1 to 21, with higher scores representing greater severity and 2.52 as minimal clinically important differences.
Change of total and sub-score of Overactive Bladder Questionnaire short form (OAB-q SF) from baseline | week 4，week 8, week 20 and week 32
  OAB-q SF is a validated questionnaire used to assess the OAB symptom bother and the health-related quality of life (HRQL) in the past 4 weeks. The domains include coping, concern, sleep and emotional interactions. The scores are transformed to a 0- to 100-point scale, with higher scores indicating severe symptoms and better HRQL.
Change of mean 24-hour pad consumption from baseline | week 4，week 8, week 20 and week 32
  The pad consumption will be documented in 3-day voiding diary.
Proportion of participants with adequate improvement assessed by Patient global impression improvement (PGI-I). | week8, week 20
  PGI-I is a global index, with only one item, used to rate the participants' subject perception on symptom improvement. Participants will describe their impression from very much better to very much worse. Adequate Improvement is defined as the response of"much better" or "very much better".
Change of mean 24-hour urgency episodes from baseline | week 4，week 8, week 20 and week 32
  The urgency episodes will be documented in 3-day voiding diary.
Change of mean 24-hour micturition episodes from baseline | week 4，week 8, week 20 and week 32
  The micturition episodes will be documented in 3-day voiding diary.

OTHER OUTCOMES:
Participants' expectations of improvement to urinary incontinence | Baseline assessment(week 0)
  Participants in the three groups will be asked: How do you expect your urinary incontinence to be in two months? Participants will choose the answer form the following options: Much better; Better; Don't know; Same; Worse；
Participants' belief that acupuncture might help | Baseline assessment(week 0) and week 4.
  In EA and SA groups, participants will be asked the question: Do you think your incontinence problem may be helped by acupuncture? Participants will choose the answer from the following options: Very ineffective; Fairly ineffective; Can't decide; Effective; Very effective；
Safety assessment | Throughout the trial
  Adverse events and severe adverse events will be recorded in case report form, whether related to interventions or not.
Blinding assessment | Within 5 minutes after either treatment at week 8
  Participants in both EA and SA groups will be asked the question: do you think you have received EA? Participants will choose the answer between the options of Yes or No.

CONTACTS AND LOCATIONS:
Overall Officials: Zhishun Liu, Study Chair — Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Locations (5):
- China (5):
  - Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - The third affiliated hospital of Beijing university of Chinese Medicine, Beijing, Beijing Municipality
  - Hengyang Hospital Affiliated to Hunan University of Chinese Medicine, Hengyang, Hunan
  - Jiangxi Provincial Hospital of traditional Chinese Medicine, Nanchang, Jiangxi
  - Yantai Hospital of Traditional Chinese Medicine, Yantai, Shandong

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underline the results reported in the article after deidentification, excluding the private information of participants.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning immediately after publication and ending 6 months following article publication
Access Criteria: Proposals should be directed to zhishunjournal@163.com. To gain access, data requestors wil need to sign a data access agreement and offer payment.

REFERENCES:
- [Derived] Sun Y, Liu Y, Chen H, Yan Y, Liu Z. Electroacupuncture for stress-predominant mixed urinary incontinence: a protocol for a three-armed randomised controlled trial. BMJ Open. 2021 Jan 7;11(1):e038452. doi: 10.1136/bmjopen-2020-038452. PMID 33414139